CLINICAL TRIAL: NCT04248244
Title: A Pilot Study to Determine the Effects of Early Palliative Care Integration on Patients With Newly Diagnosed Multiple Myeloma
Brief Title: Effects of Early Palliative Care Integration on Patients With Newly Diagnosed Multiple Myeloma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Case Comprehensive Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: CASE2A19
Record Dates: First submitted 2020-01-23; First posted 2020-01-30 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — Palliative Care; 4-amino-4'-hydroxylaminodiphenylsulfone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Early Palliative Care Integration (Experimental): 12 months of PC with concurrent standard treatment for MM, QOL assessments
  Interventions: Other: Palliative Care; Other: FACT-MM questionnaire; Other: HADS questionnaire

INTERVENTIONS:
Other: Palliative Care — Early PC Integration - Participants will meet with a member of the outpatient PC team, which consists of board-certified PC physicians, advance practice providers and nurse care coordinators, within three weeks of enrollment. Participants will be scheduled to meet with a PC provider at least once per month. Additional visits may be scheduled at the discretion of participants, oncologists or PC providers. All participants will receive routine oncologic care throughout the study period.
Other: FACT-MM questionnaire — FACT-MM questionnaires will be administered by a research coordinator upon enrollment and at four time points from the date of enrollment: 3 months, 6 months, 9 months and 12 months. All questionnaires will be administered in handwritten paper-based form, and while patients are in clinic. There is a +/- two-week window for completion of questionnaires to accommodate patient schedules. The assessment battery takes approximately 20 minutes to complete.
Other: HADS questionnaire — HADS questionnaires will be administered by a research coordinator upon enrollment and at four time points from the date of enrollment: 3 months, 6 months, 9 months and 12 months. All questionnaires will be administered in handwritten paper-based form, and while patients are in clinic. There is a +/- two-week window for completion of questionnaires to accommodate patient schedules. The assessment battery takes approximately 20 minutes to complete.

SUMMARY:
Multiple Myeloma (MM) is a common type of cancer involving the cells in the blood (commonly affecting bones, kidneys and blood). Although it remains incurable, MM has become a highly treatable form cancer thanks to new and improved treatment modalities. As patients deal with this disease, they often suffer from multiple symptoms that are caused by both the disease itself and the different drugs used to treat it. Research has shown that the most common symptoms patients suffer from include pain, constipation, tiredness, tingling in hands and feet, breathlessness, sadness and difficulty remembering things. These symptoms may negatively affect the quality of life of patients.

Palliative care (PC) is a type of treatment aimed at relieving symptoms and promoting the most optimal quality of life (QOL) for patients and their caregivers. Research has shown that patients with certain types of cancers, such as colon cancer and lung cancer, do better if they are seen by a PC provider early in the course of their disease. This study seeks to determine the effects of early PC involvement on participants with newly diagnosed MM

DETAILED DESCRIPTION:
This is a pilot study with a prospective cohort design, and based in the outpatient or ambulatory care setting. Each participant will be followed for 12 months.

Twenty eligible patients will be enrolled, and within eight weeks of diagnosis. Patients will meet with a member of the outpatient PC team, which consists of board-certified PC physicians, advance practice providers and nurse care coordinators, within three weeks of enrollment. Additional visits may be scheduled at the discretion of participants, oncologists or PC providers and participants will receive routine oncologic care throughout the study period.

The primary objective of this study is to obtain preliminary data on the effects of early PC involvement in a cohort of patients with newly diagnosed symptomatic MM

The secondary objectives of this study are to assess self-reported QOL, estimate the change in QOL relative to baseline, estimate number of participants with self-reported symptoms of depression and anxiety, to determine if monthly PC visits are feasible for participants, and to estimate health services utilization.

ELIGIBILITY:
Inclusion Criteria:

* Must be within eight weeks of being diagnosed with symptomatic MM based on current diagnostic criteria
* Able to read and respond to questions in English
* Have an ECOG performance status of 0, 1, 2 or 3
* Receiving oncologic care at a Cleveland Clinic facility

Exclusion Criteria:

* Have seen a PC provider in any setting (i.e., inpatient, outpatient or home-based)
* Need immediate referral to PC for hospice transition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-02-17 (Actual); Primary Completion 2022-10-26 (Actual); Study Completion 2022-10-26 (Actual)

PRIMARY OUTCOMES:
Self-reported QOL as measured by FACT-MM scores | At baseline
  Self-reported QOL as measured by FACT-MM scores
  The questionnaire is a combination of the original widely used and validated FACT-G (Functional Assessment of Cancer Therapy-General) questionnaire (27 items), and 14 MM-specific items.
  FACT-MM total scores range from 0 to 164, with FACT-G sections ranging from 0 to 108 and MM-specific section ranging from 0 to 56.
  Higher scores mean better QOL for all sections and total scores.
Self-reported QOL as measured by FACT-MM scores | 3 months
  Self-reported QOL as measured by FACT-MM scores The questionnaire is a combination of the original widely used and validated FACT-G (Functional Assessment of Cancer Therapy-General) questionnaire (27 items), and 14 MM-specific items.
  FACT-MM total scores range from 0 to 164, with FACT-G sections ranging from 0 to 108 and MM-specific section ranging from 0 to 56.
  Higher scores mean better QOL for all sections and total scores.
Self-reported QOL as measured by FACT-MM scores | 6 months
  Self-reported QOL as measured by FACT-MM scores The questionnaire is a combination of the original widely used and validated FACT-G (Functional Assessment of Cancer Therapy-General) questionnaire (27 items), and 14 MM-specific items.
  FACT-MM total scores range from 0 to 164, with FACT-G sections ranging from 0 to 108 and MM-specific section ranging from 0 to 56.
  Higher scores mean better QOL for all sections and total scores.
Self-reported QOL as measured by FACT-MM scores | 9 months
  Self-reported QOL as measured by FACT-MM scores The questionnaire is a combination of the original widely used and validated FACT-G (Functional Assessment of Cancer Therapy-General) questionnaire (27 items), and 14 MM-specific items.
  FACT-MM total scores range from 0 to 164, with FACT-G sections ranging from 0 to 108 and MM-specific section ranging from 0 to 56.
  Higher scores mean better QOL for all sections and total scores.
Self-reported QOL as measured by FACT-MM scores | 12 months
  Self-reported QOL as measured by FACT-MM scores The questionnaire is a combination of the original widely used and validated FACT-G (Functional Assessment of Cancer Therapy-General) questionnaire (27 items), and 14 MM-specific items.
  FACT-MM total scores range from 0 to 164, with FACT-G sections ranging from 0 to 108 and MM-specific section ranging from 0 to 56.
  Higher scores mean better QOL for all sections and total scores.
Change in QOL relative to baseline as measured by FACT-MM scores | 3 months, 6 months, 9 months and 12 months
  Change in QOL relative to baseline as measured by FACT-MM scores.
  The questionnaire is a combination of the original widely used and validated FACT-G (Functional Assessment of Cancer Therapy-General) questionnaire (27 items), and 14 MM-specific items.
  FACT-MM total scores range from 0 to 164, with FACT-G sections ranging from 0 to 108 and MM-specific section ranging from 0 to 56.
  Higher scores mean better QOL for all sections and total scores.
Number of participants with self-reported symptoms of depression and anxiety | At baseline
  Number of participants with self-reported symptoms of depression and anxiety as measured by HADS questionnaire. The questionnaire consists of 14 items, two subscales (depression and anxiety) of seven questions each for depression and anxiety. Each subsection has a possible score range of 0 to 21, with higher scores indicating worse outcomes. A score of greater than or equal to eight on either subscale is considered clinically significant (i.e., probable depression or anxiety).
Number of participants with self-reported symptoms of depression and anxiety | 3 months
  Number of participants with self-reported symptoms of depression and anxiety as measured by HADS questionnaire. The questionnaire consists of 14 items, two subscales (depression and anxiety) of seven questions each for depression and anxiety. Each subsection has a possible score range of 0 to 21, with higher scores indicating worse outcomes. A score of greater than or equal to eight on either subscale is considered clinically significant (i.e., probable depression or anxiety).
Number of participants with self-reported symptoms of depression and anxiety | 6 months
  Number of participants with self-reported symptoms of depression and anxiety as measured by HADS questionnaire. The questionnaire consists of 14 items, two subscales (depression and anxiety) of seven questions each for depression and anxiety. Each subsection has a possible score range of 0 to 21, with higher scores indicating worse outcomes. A score of greater than or equal to eight on either subscale is considered clinically significant (i.e., probable depression or anxiety).
Number of participants with self-reported symptoms of depression and anxiety | 9 months
  Number of participants with self-reported symptoms of depression and anxiety as measured by HADS questionnaire. The questionnaire consists of 14 items, two subscales (depression and anxiety) of seven questions each for depression and anxiety. Each subsection has a possible score range of 0 to 21, with higher scores indicating worse outcomes. A score of greater than or equal to eight on either subscale is considered clinically significant (i.e., probable depression or anxiety).
Number of participants with self-reported symptoms of depression and anxiety | 12 months
  Number of participants with self-reported symptoms of depression and anxiety as measured by HADS questionnaire. The questionnaire consists of 14 items, two subscales (depression and anxiety) of seven questions each for depression and anxiety. Each subsection has a possible score range of 0 to 21, with higher scores indicating worse outcomes. A score of greater than or equal to eight on either subscale is considered clinically significant (i.e., probable depression or anxiety).
Number of PC visits made in the first 12 months after diagnosis | At 12 months
  Feasibility of monthly PC visits as measured by the number of PC visits made in the first 12 months after diagnosis
Health services utilization as measured by number of ER visits, hospital admissions or ICU admissions | At 12 months
  Health services utilization as measured by number of ER visits, hospital admissions or ICU admissions

CONTACTS AND LOCATIONS:
Overall Officials: Renato Samala, MD, Principal Investigator — The Cleveland Clinic
Locations (1):
- Cleveland Clinic, Case Comprehensive Cancer Center, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No
Data from this pilot study will be used to design and power a larger prospective study.

REFERENCES:
- [Derived] Samala RV, Nurse DP, Chen X, Wei W, Crook JJ, Fada SD, Valent J. Effects of early palliative care integration on patients with newly diagnosed multiple myeloma. Support Care Cancer. 2024 Jun 27;32(7):468. doi: 10.1007/s00520-024-08665-2. PMID 38937310
- See also: Publication link — https://pubmed.ncbi.nlm.nih.gov/38937310/